CLINICAL TRIAL: NCT02868853
Title: Self-Monitoring Assessment in Real Time: 2-SMART
Brief Title: Self-Monitoring Assessment in Real Time
Acronym: 2-SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Academy of Nutrition and Dietetics (Other)
Responsible Party: Principal Investigator, Brie Turner-McGrievy, Principal Investigator, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00055836
Record Dates: First submitted 2016-07-18; First posted 2016-08-16 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Obesity
Keywords: diet; weight loss; tracking; mobile; calories
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Photo App (Experimental): Participants in this group will receive podcasts twice weekly in conjunction with using a mobile dietary tracking application(Photo App). This Photo App allows participants to track meals by taking photos.
  Interventions: Behavioral: Photo App; Behavioral: Podcasts
- Diet App (Active Comparator): Participants in this group will receive podcasts twice weekly in conjunction with an app (Diet App) to track their diet by entering in foods and beverages consumed.
  Interventions: Behavioral: Diet App; Behavioral: Podcasts

INTERVENTIONS:
Behavioral: Photo App — Use of a mobile photo app that takes pictures of foods consumed and allows users to share these pictures with other members of the study in order to receive feedback.
  Arms: Photo App
Behavioral: Diet App — Use of a mobile diet app that allows users to track all foods and beverages consumed in order to calculate the calories consumed each day.
  Arms: Diet App
Behavioral: Podcasts — Listen to 2 podcasts per week about healthy eating and exercise.

SUMMARY:
The purpose of the study is to test the effectiveness of two different methods of mobile dietary self-monitoring for weight loss. Both of these interventions will provide weight loss information through twice weekly audio podcasts. In addition to the podcasts, participants will be asked to track their diet using an assigned mobile applications (for their smartphone), which will be randomly assigned.

DETAILED DESCRIPTION:
This study will include an intensive phase for 6 weeks and a follow-up phase that will occur through the final 6 months of the study. Participants will attend one 1-hour orientation meeting at the beginning of the study and a 2-hour baseline assessment and training meeting. A final assessment will be conducted at the end of 6 weeks with a follow-up assessment at 6 months. Everyone in the study will be asked to listen to 2 podcasts per week. Each of the podcasts will take about 15-20 minutes to listen to and so participants should expect to spend 30-40 minutes each week listening to podcasts. Participants also will be randomized to track diet with one of the two mobile dietary tracking applications that will be used in the study. Participants will be encouraged to monitor their exercise and body weight.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 18-65 years old
* Own and use a smartphone and/or a tablet with a data plan that is apple of Android compatible
* BMI must be between 25-49.9 kg/m2
* Must be willing to reduce caloric intake and increase physical activity
* Not currently participating in a weight loss study or has been in a weight loss study that involved podcasts or diet apps

Exclusion Criteria:

* Over the age of 65 years old
* Currently participating in a weight loss program
* Has lost more than 10 pounds in the past 6 months
* Diagnosed with stroke or heart attack
* Diagnosed with diabetes that is controlled using medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Number of days diet is self-monitored | 6 months
  Assess the total number of days food is recorded via assigned app over the 6-week study and then assess follow-up at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Brie McGrievy, PhD, MS, RD, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dunn CG, Turner-McGrievy GM, Wilcox S, Hutto B. Dietary Self-Monitoring Through Calorie Tracking but Not Through a Digital Photography App Is Associated with Significant Weight Loss: The 2SMART Pilot Study-A 6-Month Randomized Trial. J Acad Nutr Diet. 2019 Sep;119(9):1525-1532. doi: 10.1016/j.jand.2019.03.013. Epub 2019 May 30. PMID 31155474
- [Derived] Turner-McGrievy GM, Dunn CG, Wilcox S, Boutte AK, Hutto B, Hoover A, Muth E. Defining Adherence to Mobile Dietary Self-Monitoring and Assessing Tracking Over Time: Tracking at Least Two Eating Occasions per Day Is Best Marker of Adherence within Two Different Mobile Health Randomized Weight Loss Interventions. J Acad Nutr Diet. 2019 Sep;119(9):1516-1524. doi: 10.1016/j.jand.2019.03.012. Epub 2019 May 30. PMID 31155473